CLINICAL TRIAL: NCT02819596
Title: MEDI4736 Combinations in Metastatic Renal Cell Carcinoma
Acronym: CALYPSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Vall d'Hebron Institute of Oncology (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010580QM
Record Dates: First submitted 2016-02-22; First posted 2016-06-30 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Renal Clear Cell Carcinoma; Renal Papillary Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Savolitinib (Experimental): 600 mg of Savolitinib monotherapy will administered once a day until study completion or withdrawal
  Interventions: Drug: Savolitinib
- MEDI4736 (Experimental): 1500 mg MEDI4736 will be administered every 4 weeks until study completion or withdrawal
  Interventions: Drug: MEDI4736
- Savolitinib and MEDI4736 (Experimental): Savolitinib and MEDI4736 will be administered at the Recommended Phase 2 dose ascertained in the phase Ib.
  Interventions: Drug: Savolitinib; Drug: MEDI4736
- Tremelimumab and MEDI4736 (Experimental): Subjects will receive 75 mg of Tremelimumab and 1500 mg medi4736 every 4 weeks for the first four cycles, then 750 mg MEDI4736 every 4 weeks until study completion or withdrawal.
  Interventions: Drug: MEDI4736; Drug: Tremelimumab

INTERVENTIONS:
Drug: Savolitinib
  Other Names: Volitinib; AZD6094
  Arms: Savolitinib; Savolitinib and MEDI4736
Drug: MEDI4736
  Other Names: Durvalumab
  Arms: MEDI4736; Savolitinib and MEDI4736; Tremelimumab and MEDI4736
Drug: Tremelimumab
  Arms: Tremelimumab and MEDI4736

SUMMARY:
This study is being carried out to see if the drugs MEDI4736, Savolitinib and Tremelimumab can be used alone or in combination to reduce the size of tumours in patients with kidney cancer.

The drugs being tested in this study have an anti-tumour effect and have been tested in pre-clinical and human studies before. MEDI4736 and tremelimumab work with the immune system to help the body fight against tumour cells with immune cells. Savolitinib works to correct a faulty signal which causes tumour growth.

If a patient is eligible for the study and decides to take part, they will be enrolled into one of 3 stages of the study.

* First stage [CLOSED TO RECRUITMENT]: aims to find the optimal dose of MEDI4736+savolitinib.
* Second stage [CLOSED TO RECRUITMENT]: patients with papillary cell cancer will be treated with MEDI4736+savolitinib. Patients with clear cell cancer will be randomised to one of four treatment arms and receive MEDI4736, savolitinib, MEDI4736+savolitinib, or MEDI4736+tremelimumab.
* Third stage [NOT YET OPEN TO RECRUITMENT]: patients will be tested for biomarkers before enrolment, and depending on the results will be allocated to one of 2 treatments (MEDI4736 alone or MEDI4736+tremelimumab) to see if certain biomarkers are linked to drug efficacy.

DETAILED DESCRIPTION:
This study is being carried out to see if the drugs MEDI4736, Savolitinib and Tremelimumab can be used alone or in combination to reduce the size of tumours in patients with kidney cancer.

The drugs being tested in this study have an anti-tumour effect and have been tested in pre-clinical and human studies before. MEDI4736 and tremelimumab work with the immune system to help the body fight against tumour cells with immune cells. Savolitinib works to correct a faulty signal which causes tumour growth.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performing any protocol-related procedures, including study specific screening procedures.
2. Age ≥ 18 years at the time of registration/enrolment.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥12 weeks
5. Histologically confirmed advanced (not amenable to curative surgery or radiation therapy) or metastatic (stage IV) renal cell cancer with a component of either clear cell cancer or papillary cancer. Patients with a component of both must be enrolled into the cohort with the predominant tumour type.

   1. Clear cell renal cancer patients must have experienced progressive disease after exposure to Vascular Endothelial growth rate (VEGF) targeted therapy.
   2. Sarcomatoid cell renal cancer patients must have experienced progressive disease after exposure to VEGF targeted therapy.
   3. Papillary cell renal cancer patients must be considered to be VEGF treatment naive or treatment refractory to be eligible.
6. Evidence of measurable disease as per RECIST v1.1 (i.e., ≥1 malignant tumour mass that can be accurately measured in at least 1 dimension ≥ 20 mm with conventional computerized tomography CT Scan or Magnetic Resonance Imaging (MRI), or ≥10 mm with spiral CT scan using a 5 mm or smaller contiguous reconstruction algorithm). Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable.
7. Adequate normal organ, marrow and coagulation function as defined by the following criteria:
8. Representative formalin-fixed paraffin-embedded (FFPE) tumour block with an associated anonymised pathology report must be available for central testing and determined to be evaluable for tumour assessment of PD-L1 and Met. PD-L1 and Met related testing will be required prior to study entry only for the biomarker enrichment phase of the trial. (every effort should be made to obtain FFPE blocks however unstained fresh tissue slides and core needle biopsies will suffice).
9. Patients with known tumour thrombus or deep vein thrombosis (DVT) are eligible if stable on low molecular weight heparin (LMWH) for ≥ 4 weeks.
10. Negative serum or urine pregnancy test within 2 weeks prior to the first dose of IMP (for female patients of childbearing potential only).
11. Agreement to use adequate contraceptive measures (Section 6.18).
12. Ability to swallow and retain oral medications.
13. Willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product within 28 days prior to enrolment in the study.
2. Any previous treatment with an anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody (including MEDI4736), CD137 agonists, c-MET inhibitors or pathway-targeting agents, or CTLA-4. Patients with limited c-MET inhibitor exposure must be discussed with the study medical monitor.
3. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) within 2 weeks or five half-lives of the anti-cancer therapy prior to the first dose of study drug, or radical radiotherapy within 4 weeks prior to the first dose of study drug.
4. Patients receiving strong inducers of CYP3A4, strong inhibitors of CYP3A4 or CYP1A2 or CYP3A4 substrates which have a narrow therapeutic range within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort) are excluded from enrolment in the study (see Appendix I).
5. Currently receiving treatment with therapeutic doses of warfarin sodium. LMWH is allowed.
6. Current or prior use of immunosuppressive medication within 21 days before the first dose of MEDI4736 or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
7. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL] -2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.
8. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving MEDI4736 or tremelimumab or anticipation that such a live, attenuated vaccine will be required during the study.
9. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
10. History of another primary malignancy other than renal cell carcinoma within 3 years prior to Cycle 1, Day 1 with the exception of:

    1. Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of study drug and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease e.g. cervical cancer in situ or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA <10ng/mL undergoing active surveillance and treatment naive). Patients on surveillance for low risk prostate cancer are also eligible - please discuss with medical monitor.
11. Mean resting QT interval corrected for heart rate (QTc) >470ms for women and >450ms for men calculated from triplicate electrocardiograms (ECGs) using Fridericia's correction.
12. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
13. Any unresolved toxicity of CTCAE grade >2 from previous anti-cancer therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the IMP may be included e.g. hearing loss, peripheral neuropathy etc.
14. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
15. Active or prior documented autoimmune disease within the past 2 years including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible for this study.
16. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or history of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
17. History of primary immunodeficiency
18. History of allogeneic prior allogeneic stem cell or solid organ transplant
19. History of hypersensitivity to MEDI4736, tremelimumab, or any excipient or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
20. History of hypersensitivity to savolitinib and its excipients.
21. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension (SBP>160mmHg or Diastolic blood pressure >100mmHg, patients with values above these levels must have their blood pressure controlled with medication prior to starting treatment), unstable angina pectoris, cardiac arrhythmia, or any factors that increase the risk of QTc prolongation, any clinically important abnormalities in rhythm, conduction or morphology of resting ECGs, active peptic ulcer disease or gastritis, Type I diabetes mellitus, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
22. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded.
23. Major surgical procedure within 4 weeks prior to enrolment, minor surgical procedure within 7 days of enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
24. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).
25. Active tuberculosis or known history of previous clinical diagnosis of tuberculosis.
26. History of leptomeningeal carcinomatosis
27. Female subjects who are pregnant or breast-feeding
28. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Identify Dose Limiting Toxicity -Phase Ib | 6 months
  The endpoint of this objective is to identify Dose-Limiting Toxicity that occurs during the DLT assessment phase and is almost certainty/probably dose related and drug related .Toxicity that is clearly and directly related to the primary disease or another aetiology is excluded from this definition.
Overall response (OR) in patients with metastatic clear cell renal cancer | 18 months
  Overall response rate based on RECIST V1.1 measurements taken at baseline, week 4 and every 8 weeks until disease progression
Overall response (OR) in patients with metastatic Papillary cell renal cancer | 18 months
  Overall response rate based on RECIST V1.1 measurements taken at baseline, week 4 and every 8 weeks until disease progression
Overall response (OR)in patients with metastatic renal cell cancer -Biomarker enrichment phase | 11 months
  Overall response rate based on RECIST v1.1 measurements taken at baseline, week 4 and every 8 weeks until disease progression

SECONDARY OUTCOMES:
De-escalation phase - PK-Cmax measurement | 14 months
  Measurement of Cmax for MEDI4736 and savolitinib
De-escalation phase - PK-Tmax measurement | 14 months
  Measurement of tmax for MEDI4736 and savolitinib
De-escalation phase -PK AUC (0-t) measurement | 14 months
  Measurement of AUC(0-t)for MEDI4736 and savolitinib
De-escalation phase - PK AUCs measurement | 14 months
  Measurement of AUCs for MEDI4736 and savolitinib
De-escalation phase -PK Css measurement | 14 months
  Measurement of Css max for MEDI4736 and savolitinib
De-escalation phase -PK Css min measurement | 14 months
  Measurement of Css min. for MEDI4736 and savolitinib
Expansion Phase (IIa) -Identify Progression free survival (PFS) | 18 months
  PFS defined as the time from the date of randomisation/enrolment to the date of first documented tumour progression (RECIST V1.1) or death from any cause , whichever occurs first
Expansion Phase (IIa) -Identify overall Survival (OS) | 18 months
  OS defined as the time from study entry to death from any cause. All deaths will be included whether they occur on study or following treatment discontinuation. For patients who have not died, overall survival will be censored at the date of last contact
Expansion Phase (IIa) -Identify duration of response | 18 months
  Duration of response defined as the time from first documentation of CR or PR to disease progression (RECIST v1.1) or death from any cause, whichever occurs first.
Biomarker positive patient analysis | 11 months
  Patients that have test positive for C-met or PD-L1 alterations;OS defined as the time from study entry to death from any cause.All deaths will be included whether they occur on study or following treatment discontinuation. For patients who have not died, overall survival will be censored at the date of last contact
Biomarker positive patient analysis | 11 months
  Patients that have test positive for C-met or PD-L1 alterations; PFS defined as the time from the date of registration to the date of the first documented tumour progression as per RECIST V1.1 or death from any cause , whichever occurs first
Expansion Phase (IIa) -Best Response | 18 months
  Best response after 24 weeks of treatment as assessed by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Powles, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Powles T et al. CALYPSO: A three-arm randomized phase II study of durvalumab alone or with savolitinib or tremelimumab in previously treated advanced clear cell renal cancer. Journal of Clinical Oncology 40, no. 17_suppl (June 10, 2022) LBA4503-LBA4503
- [Result] Suarez C, Larkin JMG, Patel P, Valderrama BP, Rodriguez-Vida A, Glen H, Thistlethwaite F, Ralph C, Srinivasan G, Mendez-Vidal MJ, Hartmaier R, Markovets A, Prendergast A, Szabados B, Mousa K, Powles T. Phase II Study Investigating the Safety and Efficacy of Savolitinib and Durvalumab in Metastatic Papillary Renal Cancer (CALYPSO). J Clin Oncol. 2023 May 10;41(14):2493-2502. doi: 10.1200/JCO.22.01414. Epub 2023 Feb 21. PMID 36809050
- [Result] Suarez Rodriguez et al. Overall survival results for durvalumab and savolitinib in metastatic papillary renal cancer. Journal of Clinical Oncology 2020 38:6_suppl, 619-619.
- [Result] Suarez Rodriguez et al Clinical activity of durvalumab and savolitinib in MET-driven, metastatic papillary renal cancer. J Clin Oncol 39, 2021 (suppl 15; abstr 4511).